CLINICAL TRIAL: NCT02925169
Title: Shape and Dimensions of the Upper Airway in Infants Using Computed Tomography Imaging
Status: Completed | Type: Observational
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Tariq Wani, Consultant, Pediatric Anesthesia, King Fahad Medical City
Other Study IDs: H-01-R-012
Record Dates: First submitted 2016-07-16; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Child
Keywords: Subglottis, cricoid, airway shape, CT imaging
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CT Scan — CT imaging

SUMMARY:
Cricoid is considered the narrowest part with the shape of airway defined as elliptical with the subglottis as the narrowest region.

This study using imaging modality (2D CT images) is done to determine any differences in airway shape between infants and children, and to evaluate the dimensional transition between the subglottic area and the cricoid ring.

DETAILED DESCRIPTION:
Using imaging modalities (CT, MRI), the funnel-shape of the airway in children has been questioned and subglottis rather than cricoid is considered the narrowest part with the shape of airway defined as elliptical with the subglottis as the narrowest region.

This is the first study using imaging modality (2D CT images) to determine the airway shape and dimensions in neonates and infants. The purpose of this investigation was to determine any differences in airway shape between infants and children, and to evaluate the dimensional transition between the subglottic area and the cricoid ring.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants.

Exclusion Criteria:

Patients with tracheostomy, tracheo-esophageal fistulas lung collapse mediastinal masses diaphragmatic hernias chest masses intubated patients patients, preterm infants syndromic patients patients with primary lung diseases

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children less than 12 months of age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Shape of airway in neonates and infants | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Wani, MD, Principal Investigator — King Fahad Medical City
Locations (1):
- King Fahad Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wani TM, Bissonnette B, Rafiq Malik M, Hayes D Jr, Ramesh AS, Al Sohaibani M, Tobias JD. Age-based analysis of pediatric upper airway dimensions using computed tomography imaging. Pediatr Pulmonol. 2016 Mar;51(3):267-71. doi: 10.1002/ppul.23232. Epub 2015 Jun 17. PMID 26083203
- [Background] Sellars I, Keen EN. Laryngeal growth in infancy. J Laryngol Otol. 1990 Aug;104(8):622-5. doi: 10.1017/s0022215100113416. PMID 2230557
- [Background] Litman RS, Weissend EE, Shibata D, Westesson PL. Developmental changes of laryngeal dimensions in unparalyzed, sedated children. Anesthesiology. 2003 Jan;98(1):41-5. doi: 10.1097/00000542-200301000-00010. PMID 12502977